CLINICAL TRIAL: NCT04599127
Title: Mobilization With Movement as an Additional Treatment to Conventional Physical Therapy in Individuals With Shoulder Impingement Syndrome
Brief Title: The Effect of Mobilization With Movement in Individuals With Shoulder Impingement Syndrome
Acronym: SIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MWM
Record Dates: First submitted 2020-05-10; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Shoulder Impingement Syndrome; Subacromial Impingement; Subacromial Impingement Syndrome; Subacromial Pain Syndrome; Impingement Syndrome, Shoulder
Keywords: Shoulder impingement syndrome; Mobilization with movement; Conventional physical therapy; Pain intensity; Visual analogue scale; Range of motion; Inclinometer; Shoulder pain and disability index; Postural assessment software; Craniovertebral angle; Sagittal shoulder posture; Hand held dynamometer
MeSH Terms: conditions — Shoulder Impingement Syndrome; Pain; Shoulder Pain | interventions — Movement

STUDY DESIGN:
Intervention Model Description: All of the eligible participants will be divided into two groups; conventional physical therapy and conventional physical therapy plus mobilization with movement
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participant will be blinded by unknowing the randomization of the group allocation using a sealed envelope.
  The physical therapy (S) who treats the participants using mobilization with movement will be blinded by unknowing the group allocation of the participants.
  The physical therapy (E) who treats the participants using conventional physical therapy will be blinded by unknowing the group allocation because all of the participants will be treated using conventional physical therapy.
  The examiner (AH) and (FN) will be blinded by unknowing the participant group and the sequence of assessments will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization with movement (Experimental): Mobilization with movement on the shoulder abduction and external rotation
  Interventions: Other: Mobilization with movement; Other: Conventional physical therapy
- Conventional physical therapy (Placebo Comparator): Postural correction exercise and muscle strengthening of the rotator cuff muscle and surrounding muscle on the subacromial region
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Mobilization with movement — The physical therapist will adjust the active movement of the shoulder joint during the arm elevation or abduction and shoulder external rotation
  Other Names: Mulligan techniques
  Arms: Mobilization with movement
Other: Conventional physical therapy — The exercise is tailor-made and each participant will be performing some of the exercises based on the list that physical therapist prescription
  Other Names: Postural correction exercise

SUMMARY:
This study conducted to see the effect of adding mobilization with movement to conventional physical therapy to the subject with shoulder impingement syndrome. The shoulder impingement syndrome is often described as anterior lateral shoulder pain that provoked during shoulder elevation. The pain occurs during shoulder elevation and causes limited range of motion. Moreover, the patients with shoulder impingement syndrome commonly had a forward head posture and slouching shoulder. There is a theory that illustrates the mechanical factors lead to the injury of the bursa or rotator cuff tendons below the subacromial space which is highly related to the posture and scapular movement.

Various treatments for shoulder impingement syndrome including medical treatments such as anti-inflammatory drugs, subacromial decompression, and acromion resection surgery. Conventional physical therapy treatments for shoulder impingement syndrome included modalities, exercises and manual therapy. Exercise has been showed to give a significant effect to decrease the pain intensity, increasing the range of motion and shoulder function. There is evidence that supports the use of manual therapy on shoulder impingement, the recent technique introduced by Brian Mulligan is mobilization with movement. Mobilization with movement is a manual therapy technique that uses the active movement while the physical therapist applies an accessory force to align the positional fault of the joint. A previous study investigated the effect of mobilization with movement that uses the mobilization with movement in shoulder impingement syndrome showed different outcomes in the measurement of pain intensity and shoulder range of motion. As the posture may be related to shoulder impingement syndrome, this research will measure the cervical posture, shoulder posture, and muscle strength.

Therefore, the purposes of this study will be to compare the effects of conventional physical therapy treatments and the conventional therapy treatments plus the mobilization with movement on pain intensity, shoulder range of motion, cervical and shoulder posture, shoulder muscle strength and shoulder function. The study hypothesis was that mobilization with movement is more effective in improving the investigated outcomes in individuals with shoulder impingement syndrome than the conventional physical therapy.

DETAILED DESCRIPTION:
Shoulder impingement syndrome causes positional fault of the subacromial and soft tissues below the subacromial space. This condition leads to the wrong biomechanics of precise ball and socket kinematics creating maximum concavity compression for shoulder stability. This wrong biomechanics is resulting in the injury of tissue below the subacromial space, such as rotator cuff tendinitis, tears of rotator cuff tendons, and subacromial bursitis. The space between the acromion and humeral was small varying between nine to 14 mm. However, the subacromial space will be decreased during the arm elevation or in the abduction and external rotation position. Some of the researchers defined the shoulder impingement syndrome as the mechanical entrapment of the rotator cuff or the subacromial bursa in the subacromial space. The highest compression of the structures below the subacromial space occurs when people elevate the arm, especially during the shoulder flexion, abduction, and rotation.

The etiology of shoulder impingement syndrome is multifactorial, although a few common causes of the shoulder impingement syndrome were narrowing of the subacromial space and enlargement of the subacromial bursa or rotator cuff tendons. The mechanical factor is believed as the main cause of shoulder impingement syndrome. The postural misalignment and the movement control that makes the improper muscle activation and cause false movement times between acromion and glenoid were shown to associated with the etiology of shoulder impingement syndrome. Individu with the protracted shoulder is frequently associated with the anteriorly tilted and internally rotated of the scapula. The protracted shoulder or forward displacement of the acromion can be measured by the shoulder angle to the seventh cervical spinous process.

The humeral head position depends on the soft tissues surrounding the subacromial region. During arm elevation, the humeral head position should be at the center and adjust anterior translation along with the acromion movement to anterior and lateral. When the humeral head position is faulty or not in the center, because of the anterior inferior glenohumeral ligament cannot restrain the abnormal humeral head translation. This condition leads to decreased subacromial space and irritation to the soft tissue below the acromion which causes the impingement syndrome.

Study protocol This study will recruit shoulder patients around Jakarta city, the age between 20 and 60 years. The patients with shoulder impingement syndrome will be recruited by online brochures and leaflets.

All eligible participants will receive a clear explanation of the purposes, procedures, advantages, and possible risks of this study. Each participant will be asked to sign an informed consent after they understand and accept to participate in this study.

Based on the assessment form, the participant will be assessed by the examiner and researcher. The participants' age will be used to grouping the participants into the conventional or mobilization with the movement group. The participant will be asked to rate their pain intensity using the visual analog scale during the maximum shoulder abduction. Shoulder range of motion will be assessed using the bubble inclinometer during shoulder abduction in the standing position, internal and external rotation in the supine position with 90° shoulder abduction and 90° elbow flexion. Cervical and shoulder with the instruction to the participants to stand in their relaxed posture will be recorded by photogrammetry. Muscle strength of shoulder abductors, external rotators, and internal rotators will be assessed using the handheld dynamometer. The shoulder function will be recorded by the shoulder pain and disability index.

Conventional physical therapy For the conventional group, PT (E), who has had certified level 1 sports physical therapy from the Australian Physiotherapy Association and has had 5 years of working experience, will treat the participants with the conventional and postural correction exercise. This therapist will be blinded by unknowing the group allocation. The participants will receive the conventional intervention, the postural correction exercise, and 10 minutes rest. Then the outcome measures will be reassessed thereafter. The participants in the conventional group will receive conventional physical therapy including stretching, modality, ice, therapeutic exercise, passive mobilization, and postural correction exercise. The conventional physical therapy is adjustable or tailor-made depending on the patient's specific conditions. Therapeutic exercise has a wide variety of types and modes of exercise. The postural correction exercises consist of rotator cuff muscle strengthening with eccentric-concentric, scapular stabilization exercise, and postural awareness. In addition, these exercises include motor control therapeutic exercise for the relearn process and motor control of the correct posture to change the participant's behavior.

Mobilization with movement For the mobilization with movement group, PT (S) will know the code to treat the participants using the conventional or mobilization with movement protocol. Moreover, this therapist will apply the mobilization with movement technique. The participants will receive the conventional intervention, the postural correction exercise, and the mobilization with movement. Then the outcome measures will be reassessed thereafter. The directions of mobilization with movement are a posterolateral glide when the participants raise their arm to perform shoulder abduction until the overhead movement. The therapist will place one hand on the participant's scapula to stabilize movement while placing the thenar eminence of the other hand on the medial of the humeral head. The treatment belt will be placed on the participant's shoulder on top of the PT (S)'s hand. The therapist will provide sustained posterolateral and inferior glide while the participants will be asked to move the shoulder freely in the pain-free angle. PT (S)'s hands will move along with the movement to sustain the glide along the treatment plane with upward rotation of the scapula. The mobilization with movement dose will be 3 sets of 10 repetitions with rest interval 30 seconds between sets, twice a week for 4 weeks.

Sample size calculation will be performed using the formula for the test of the difference between 2 independent means.

According to the G*power 3.1.9.2 program calculation, the total of this study equals 20 subjects. Based on the previous study using the shoulder pain and disability index to measure the shoulder function, in the study of comparing the immediate effects of mobilization with movement and sham techniques. The mean (standard deviation) between group post-intervention for the mobilization with movement group was 4.6 (5.0) and that for the sham group was 0.4 (1.1). In this proposed study, the investigators need an equal number of participants per group; therefore, the drop out the calculation of 20% of the total participants (n = 1/1-20%). Therefore, after the ethical approval, the researcher will collect data from 24 shoulder impingement syndrome patients (12 subjects on the conventional group and 12 subjects on the mobilization with movement group).

Statistical Analysis Data will be analyzed using SPSS version 23. The statistical significance level is set at a p-value < 0.05.

* Shapiro-Wilk will be used to examine the distribution of the data
* Descriptive statistics for demographic data, mean and standard deviation for continuous, cumulative frequency for categorical, and median for ordinal variables, will be calculated.
* Two-way mixed-design ANOVA (two group x four-time) for parametric data. If the data are significant the post hoc analysis will be performed using Bonferroni.
* Friedman tests if the data are not normally distributed.

ELIGIBILITY:
Inclusion Criteria:

* Anterior and/or lateral shoulder pain (between the acromion and glenoid)
* Score 4 - 7 cm on the 0 - 10 visual analog scale
* Experienced shoulder pain at least 3 months
* Positive combination 2 of 3 impingement test (painful arc, empty can, and external rotation test)
* Negative at least one of rotator cuff test (isometric infraspinatus and subscapularis muscle test)

Exclusion Criteria:

* History of shoulder, cervical, or thoracic surgery
* History of neurological conditions (stroke, brachial plexus injury)
* Postural deformity and musculoskeletal condition that affects the shoulder movement
* History of shoulder major trauma on the affected side (fracture, dislocation, tendon rupture and/or lateral torn)
* Having bilateral shoulder impingement syndrome
* Recently using muscle relaxants, pain killer, or corticosteroid injection
* Ligamentous laxity based on positive sulcus sign
* Numbness or tingling in upper extremity
* Systemic illness or widespread pain
* Rheumatic disease
* Having malfunction of the rotator cuff (e.g. cannot perform at all)
* Having a passive limitation due to adhesive capsulitis
* Positive of scapular retraction test

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Pain intensity change between time | Baseline, at the week 1, week 2, week 3, and week 4
  Visual analogue scale, 0 mean no pain at all until 10 scale mean the worst pain
Shoulder function change between time | Baseline, at the week 2, and week 4
  Shoulder pain and disability index, this index is consist of 13 items with 0 score mean no pain and 10 score mean the worst pain imaginable, the scoring calculation is that the total score / 130 x 100 = ___%

SECONDARY OUTCOMES:
Range of motion change between time | Baseline, at week 1, week 2, week 3, and week 4
  Inclinometer, measure the joint range of motion with 0 degree mean no motion at all and 180 degree is the maximum range for the shoulder abduction motion
Muscle strength change between time | Baseline, at week 2 and week 4
  Hand held dynamometer, measure the peak isometric force with 0 score mean there is no contraction of the muscle, the maximum isometric force of each individual can be vary from 1 kgf to the limit
Postural assessment change between time | Baseline, at week 2 and week 4
  Craniovertebral angle and sagittal shoulder posture, measures using the postural assessment software (PAS) to see the degree of craniovertebral angle and sagittal shoulder posture angle. The degree varying on each individual, the smallest craniovertebral angle mean that the person is more forward head and the smallest sagittal shoulder posture mean that the person is more slouchy.

CONTACTS AND LOCATIONS:
Overall Officials: Wunpen Chansirinukor, Dr., Study Director — Mahidol University
Locations (1):
- Esa Unggul physical therapy clinic, Jakarta, Jakarta Barat, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
The study protocols and the participant's data record with only initial or code
Supporting Information: Study Protocol
Time Frame: The data will be available in May 2020 and will be held until two years after the data collection is done
Access Criteria: The access for the data will be shared using the Mahidol University Physical therapy e-library and anyone can get access by contacting the administrator
URL: https://www.li.mahidol.ac.th/e-databases/

REFERENCES:
- [Background] Linsell L, Dawson J, Zondervan K, Rose P, Randall T, Fitzpatrick R, Carr A. Prevalence and incidence of adults consulting for shoulder conditions in UK primary care; patterns of diagnosis and referral. Rheumatology (Oxford). 2006 Feb;45(2):215-21. doi: 10.1093/rheumatology/kei139. Epub 2005 Nov 1. PMID 16263781
- [Background] Singla D, Veqar Z, Hussain ME. Photogrammetric Assessment of Upper Body Posture Using Postural Angles: A Literature Review. J Chiropr Med. 2017 Jun;16(2):131-138. doi: 10.1016/j.jcm.2017.01.005. Epub 2017 Mar 18. PMID 28559753
- [Result] Dong W, Goost H, Lin XB, Burger C, Paul C, Wang ZL, Zhang TY, Jiang ZC, Welle K, Kabir K. Treatments for shoulder impingement syndrome: a PRISMA systematic review and network meta-analysis. Medicine (Baltimore). 2015 Mar;94(10):e510. doi: 10.1097/MD.0000000000000510. PMID 25761173
- [Result] Ho CY, Sole G, Munn J. The effectiveness of manual therapy in the management of musculoskeletal disorders of the shoulder: a systematic review. Man Ther. 2009 Oct;14(5):463-74. doi: 10.1016/j.math.2009.03.008. Epub 2009 May 21. PMID 19467911
- [Result] Teys P, Bisset L, Vicenzino B. The initial effects of a Mulligan's mobilization with movement technique on range of movement and pressure pain threshold in pain-limited shoulders. Man Ther. 2008 Feb;13(1):37-42. doi: 10.1016/j.math.2006.07.011. Epub 2006 Oct 27. PMID 17070090
- [Result] Senbursa G, Baltaci G, Atay A. Comparison of conservative treatment with and without manual physical therapy for patients with shoulder impingement syndrome: a prospective, randomized clinical trial. Knee Surg Sports Traumatol Arthrosc. 2007 Jul;15(7):915-21. doi: 10.1007/s00167-007-0288-x. Epub 2007 Feb 28. PMID 17333123
- [Result] DeSantis L, Hasson SM. Use of Mobilization with Movement in the Treatment of a Patient with Subacromial Impingement: A Case Report. J Man Manip Ther. 2006 Apr 18;14(2):77-87.
- [Result] Delgado-Gil JA, Prado-Robles E, Rodrigues-de-Souza DP, Cleland JA, Fernandez-de-las-Penas C, Alburquerque-Sendin F. Effects of mobilization with movement on pain and range of motion in patients with unilateral shoulder impingement syndrome: a randomized controlled trial. J Manipulative Physiol Ther. 2015 May;38(4):245-52. doi: 10.1016/j.jmpt.2014.12.008. Epub 2015 Apr 30. PMID 25936465
- [Result] Guimaraes JF, Salvini TF, Siqueira AL Jr, Ribeiro IL, Camargo PR, Alburquerque-Sendin F. Immediate Effects of Mobilization With Movement vs Sham Technique on Range of Motion, Strength, and Function in Patients With Shoulder Impingement Syndrome: Randomized Clinical Trial. J Manipulative Physiol Ther. 2016 Nov-Dec;39(9):605-615. doi: 10.1016/j.jmpt.2016.08.001. Epub 2016 Nov 6. PMID 27829501
- [Result] Kachingwe AF, Phillips B, Sletten E, Plunkett SW. Comparison of manual therapy techniques with therapeutic exercise in the treatment of shoulder impingement: a randomized controlled pilot clinical trial. J Man Manip Ther. 2008;16(4):238-47. doi: 10.1179/106698108790818314. PMID 19771196
- [Result] Menek B, Tarakci D, Algun ZC. The effect of Mulligan mobilization on pain and life quality of patients with Rotator cuff syndrome: A randomized controlled trial. J Back Musculoskelet Rehabil. 2019;32(1):171-178. doi: 10.3233/BMR-181230. PMID 30248039
- [Result] Surenkok O, Aytar A, Baltaci G. Acute effects of scapular mobilization in shoulder dysfunction: a double-blind randomized placebo-controlled trial. J Sport Rehabil. 2009 Nov;18(4):493-501. doi: 10.1123/jsr.18.4.493. PMID 20108851
- [Result] Ludewig PM, Cook TM. Alterations in shoulder kinematics and associated muscle activity in people with symptoms of shoulder impingement. Phys Ther. 2000 Mar;80(3):276-91. PMID 10696154
- [Result] Seitz AL, Podlecki LA, Melton ER, Uhl TL. NEUROMUSCULAR ADAPTIONS FOLLOWING A DAILY STRENGTHENING EXERCISE IN INDIVIDUALS WITH ROTATOR CUFF RELATED SHOULDER PAIN: A PILOT CASE-CONTROL STUDY. Int J Sports Phys Ther. 2019 Feb;14(1):74-87. PMID 30746294
- [Result] Ellenbecker TS, Cools A. Rehabilitation of shoulder impingement syndrome and rotator cuff injuries: an evidence-based review. Br J Sports Med. 2010 Apr;44(5):319-27. doi: 10.1136/bjsm.2009.058875. PMID 20371557
- [Result] Moezy A, Sepehrifar S, Solaymani Dodaran M. The effects of scapular stabilization based exercise therapy on pain, posture, flexibility and shoulder mobility in patients with shoulder impingement syndrome: a controlled randomized clinical trial. Med J Islam Repub Iran. 2014 Aug 27;28:87. eCollection 2014. PMID 25664288
- [Result] Satpute KH, Bhandari P, Hall T. Efficacy of Hand Behind Back Mobilization With Movement for Acute Shoulder Pain and Movement Impairment: A Randomized Controlled Trial. J Manipulative Physiol Ther. 2015 Jun;38(5):324-34. doi: 10.1016/j.jmpt.2015.04.003. Epub 2015 Jun 20. PMID 26099206
- [Result] Brudvig TJ, Kulkarni H, Shah S. The effect of therapeutic exercise and mobilization on patients with shoulder dysfunction : a systematic review with meta-analysis. J Orthop Sports Phys Ther. 2011 Oct;41(10):734-48. doi: 10.2519/jospt.2011.3440. Epub 2011 Sep 4. PMID 21891875
- Available data/document: Study Protocol: MU-CIRB 2019/206.06.08 — https://sp.mahidol.ac.th/eng/contact-mucirb.html — The data can be accessed by using the ethics committee of Mahidol University Central Institutional Review Board to see the ethics approval protocols with the code: MU-CIRB 2019/206.06.08 or using the email to feypqbd@yahoo.com

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-02-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT04599127/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT04599127/ICF_001.pdf